CLINICAL TRIAL: NCT06376344
Title: The Effect of Myofascial Release Using a Tennis Ball on Balance and Quality of Life in Cancer Patients With Peripheral Neuropathy: a Randomized Controlled Trial.
Brief Title: The Effect of Tennis Ball on Balance and Quality of Life in Cancer Patients With Neuropathy.
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Ülkü Saygılı, Assist. Prof, Selcuk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 16.04.24
Record Dates: First submitted 2024-04-16; First posted 2024-04-19 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Cancer; Neuropathy; Therapy-Associated Cancer
Keywords: Cancer pain; Neuropathy pain; Tenis ball; Myofascial release
MeSH Terms: conditions — Neoplasms; Neoplasms, Second Primary; Cancer Pain | interventions — Myofascial Release Therapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study (Experimental)
  Interventions: Other: myofascial release with tennis ball
- Control (No Intervention)

INTERVENTIONS:
Other: myofascial release with tennis ball — Movement of the Tennis Ball on the Sole of the Foot: The tennis ball is moved under the foot by back and forth movements and by applying pressure. The aim is to briefly keep the pressure of the ball on the body and the stress indicated by the massage on.
  Arms: Study

SUMMARY:
This research; It was aimed to evaluate the effect of myofascial release using a tennis ball on balance and quality of life in cancer patients who developed peripheral neuropathy.

ELIGIBILITY:
Inclusion Criteria:

* Complaints of peripheral neuropathy among patients who have completed the standard chemotherapy treatment protocol due to colorectal cancer, entered the follow-up process and come to the outpatient clinic for routine control.
* Registered to Selçuk University Faculty of Medicine Hospital Medical Oncology Polyclinic
* Karnofsky Performance Scale must be 80 or above
* Over 25 years old, under 65 years old
* Presence of grade 2 or higher peripheral neuropathy,
* Being conscious and cooperative
* Verbal and written approval to participate in the study after an explanation about the study is made.

Exclusion Criteria:

* Having any skin sensitivity on hands and feet before
* Refused to participate in the study after making a statement about the study
* Development of peripheral neuropathy due to reasons other than chemotherapy [tumor compression, nutritional disorders, infections or major systemic disease (diabetes mellitus, etc.)]
* Bone or spine metastases

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-04-28 (Estimated); Primary Completion 2024-06-10 (Estimated); Study Completion 2024-07-10 (Estimated)

PRIMARY OUTCOMES:
EORTC QLQ C-30- CIPN20 Scale | 10 minutes
  The patients' quality of life will be evaluated with the EORTC QLQ-C30, which was developed by EORTC for cancer patients and is widely used all over the world. The first 28 of the scale, which consists of three subheadings and 30 questions, namely functional difficulties, symptom control and general well-being, are four-point Likert type, and the answers are given as "Not at all", "Somewhat", "2", Somewhat "3", Very "4". is evaluated. In the 29th and 30th questions of the scale, the patient is asked to evaluate his/her general well-being by using a linear analog scale and giving a value from 1 to 7 ("1" is very bad and "7" is excellent). Functional scale: physical function (questions 1-5), role function (questions 6 and 7), emotional function (questions 21-24), cognitive function (questions 20 and 25) and social function (questions 26 and 27). )consists of subgroups
One Leg Standing Test | 30 seconds
  During the test, the participant is asked to cross his arms in front of his body and lift one leg without touching the support leg. Initially, his eyes are open. The eyes are fixed in the direction of the head, the participant is asked to close his eyes and is expected to maintain his balance for 30 seconds.
Lateral Reach Test | 5 minutes
  In the lateral reach test, the participant is asked to turn his back to the wall, stand close to it but not touch it, and keep his arm close to the wall by abducting it at 90 degrees
Pain Assessment | 1 minutes
  Pain will be assessed with the Visual Analog Scale (VAS) [20]. Patients are explained that the number "0" on a 10 cm horizontal line means no pain, and the number "10" means "unbearable pain
Pressure Pain Threshold Assessment | 5 minutes
  In quantitative pain threshold measurement, a 1 cm2 surface algometer will be used to measure the pressure pain threshold. The algometer is positioned upright, the pressure is increased to 1kg/cm2 at the painful point every three seconds, and the measurements are repeated 3 times with a 30-second rest period in between. The average of 3 measurements is used for analysis.
Two Point Discrimination | 10 minutes
  Participants will be evaluated in a sitting position with eyes closed using an aesthesiometer (Instrument Company, Lafayette, IN, USA). Evaluation will be made from the trans-metatarsal area, middle of the foot and middle of the heel. It will start from the interval where two points can be easily distinguished. The distance between two points will be reduced in 1 mm intervals until the two points are felt as a single point.

CONTACTS AND LOCATIONS:
Locations (1):
- ülkü Saygili Düzova, Selçuklu, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided